CLINICAL TRIAL: NCT06015867
Title: Effect of Sourdough Bread Consumption on Postprandial Responses, Appetite Regulation and Energy Intake at the Subsequent Meal (SPAR Study)
Brief Title: Effect of Sourdough Bread Consumption on Postprandial Responses, Appetite Regulation and Energy Intake
Acronym: SPAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Kristin Verbeke, Full professor, KU Leuven
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: S64824 - B3222020000339
Record Dates: First submitted 2023-08-22; First posted 2023-08-29 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Appetite; Satiety; Energy Intake; Glucose Response; Insulin Response; Gastric Emptying
MeSH Terms: interventions — Diet Therapy; Yeast, Dried

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Bread: Wholemeal Yeast Bread (Active Comparator): Wholemeal bread, containing mainly of wholemeal flour, water and bakers' yeast will be used as the control test bread.
  Interventions: Dietary Supplement: Dietary Intervention with Wholemeal Bread with Yeast; Dietary Supplement: Dietary Intervention with Wholemeal Sourdough Bread
- Wholemeal Sourdough Bread (Active Comparator): Wholemeal sourdough bread, containing mainly of wholemeal flour, water and added sourdough co-culture (consisting of W.anom.+ C.crust strain).
  Interventions: Dietary Supplement: Dietary Intervention with Wholemeal Bread with Yeast; Dietary Supplement: Dietary Intervention with Wholemeal Sourdough Bread

INTERVENTIONS:
Dietary Supplement: Dietary Intervention with Wholemeal Bread with Yeast — Single administration of 150g wholemeal long-time processed bread with baker's yeast, with no lactic acid (control).
Dietary Supplement: Dietary Intervention with Wholemeal Sourdough Bread — Single administration of 150g wholemeal long-time processed sourdough bread (with alternative lactic acid bacteria and yeast) high in lactic acid concentration.

SUMMARY:
During this project the effect of yeast bread and sourdough breads consumption on satiety, energy intake at subsequent meal and postprandial metabolic responses, will be investigated.

DETAILED DESCRIPTION:
The primary aim of this study will be to evaluate the impact of an alternative starter culture that produces high levels of lactic acid on appetite regulation (subjective satiety and energy intake at the subsequent meal). The second aim will be to identify mechanistic parameters that may explain the observed effects, including glycaemic and insulin response, and gastric emptying rate. In addition, habitual physical activity levels, and mood and stress levels of the subjects will be evaluated as potential covariates of appetite regulation.

It is hypothesized that:

Sourdough breads fermented with the alternative starter culture that produce high concentrations of lactic acid will reduce glucose response via lower starch digestibility and/or slower gastric emptying rate. The reduced glycaemic response will lead to higher satiety and lower energy intake at the subsequent meal (more than 10%).

ELIGIBILITY:
Inclusion Criteria:

* Female and male participants
* age range 18 - 50
* BMI range 18.5 - 25.0 kg/m2 at screening visit
* Regular eating pattern (3 meals per day on at least 5 days per week)
* Stable body weight for the last 6 months

Exclusion Criteria:

* Currently smoking (has smoked in the last 28 days) or willingness to smoke during the study period
* Pregnancy, lactation or wish to become pregnant during the study period
* Family history of diabetes
* Previous or current gastrointestinal or endocrine disorders
* Previous or current substance/alcohol dependence or abuse (> 2 units per day/14 units per week)
* Coeliac disease or gluten sensitivity
* Use of pre- or probiotics within one month preceding the study
* Use of antibiotics within 3 months preceding the study
* Excessive concern about eating habits or body weight as evidenced from scores < 18 on the restraint and disinhibition subscales of the Three-Factor Eating Questionnaire (Stunkard & Messick, 1985)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-04-28 (Actual); Study Completion 2024-04-28 (Actual)

PRIMARY OUTCOMES:
Appetite measurements | During test day 1 (up to 4 hours)
  Appetite in response to test meal, will be measured using 100 millimeter (mm) Visual Analogue Scales (VAS), with 0 being the minimum value (not at all) and 100 being the maximum value (extremely).
  Measurements will be taken: before eating (i.e. 0 minute) and at respective time points after completion of test meal (I.e. 15, 30, 45, 60, 75, 90, 105, 120, 135, 150, 165, 180, 195, 210, 225, 240 minutes).
Appetite measurements | During test day 2 (up to 4 hours)
  Appetite in response to test meal, will be measured using 100 millimeter (mm) Visual Analogue Scales (VAS), with 0 being the minimum value (not at all) and 100 being the maximum value (extremely).
  Measurements will be taken: before eating (i.e. 0 minute) and at respective time points after completion of test meal (I.e. 15, 30, 45, 60, 75, 90, 105, 120, 135, 150, 165, 180, 195, 210, 225, 240 minutes).
Food intake at subsequent meal | During test day 1 (240 minutes after ingestion of breakfast)
  Weighted amounts of ad-libitum food offered minus the weighted leftovers
Food intake at subsequent meal | During test day 2 (240 minutes after ingestion of breakfast)
  Weighted amounts of ad-libitum food offered minus the weighted leftovers

SECONDARY OUTCOMES:
Glucose response | During test day 1 (up to 4 hours)
  Blood glucose response will be measured through blood samples collected via placed catheter before eating and at respective time points after completion of test meal (I.e. 0, 15, 30, 45, 60, 75, 90, 105, 120, 150, 180, 210, 240 minutes)
Glucose response | During test day 2 (up to 4 hours)
  Blood glucose response will be measured through blood samples collected via placed catheter before eating and at respective time points after completion of test meal (I.e. 0, 15, 30, 45, 60, 75, 90, 105, 120, 150, 180, 210, 240 minutes)
Insulin response | During test day 1 (up to 4 hours)
  Blood C-peptide (as indicator of insulin response) will be measured through blood samples collected via placed catheter before eating and at respective time points after completion of test meal (I.e. 0, 15, 30, 45, 60, 75, 90, 105, 120, 150, 180, 210, 240 minutes)
Insulin response | During test day 2 (up to 4 hours)
  Blood C-peptide (as indicator of insulin response) will be measured through blood samples collected via placed catheter before eating and at respective time points after completion of test meal (I.e. 0, 15, 30, 45, 60, 75, 90, 105, 120, 150, 180, 210, 240 minutes)
Gastric emptying rate | During test day 1 (up to 4 hours)
  Gastric emptying rate will be measured through 13C-octanoic acid breath samples collected before eating (i.e. 0 minute) and at respective time points after completion of test meal (I.e. 15, 30, 45, 60, 75, 90, 105, 120, 135, 150, 165, 180, 195, 210, 225, 240 minutes).
Gastric emptying rate | During test day 2 (up to 4 hours)
  Gastric emptying rate will be measured through 13C-octanoic acid breath samples collected before eating (i.e. 0 minute) and at respective time points after completion of test meal (I.e. 15, 30, 45, 60, 75, 90, 105, 120, 135, 150, 165, 180, 195, 210, 225, 240 minutes).
Subjective stress ratings | During test day 1 (up to 4 hours)
  Subjective stress, will be measured using 100 millimeter (mm) Visual Analogue Scales (VAS), with with 0 being the minimum value (not at all) and 100 being the maximum value (extremely).
  Measurements will be takem: before eating (i.e. -15 minute) and at respective time points after completion of test meal (I.e. 0, 60, 120, 180, 240 minutes).
Subjective stress ratings | During test day 2 (up to 4 hours)
  Subjective stress, will be measured using 100 millimeter (mm) Visual Analogue Scales (VAS), with with 0 being the minimum value (not at all) and 100 being the maximum value (extremely).
  Measurements will be takem: before eating (i.e. -15 minute) and at respective time points after completion of test meal (I.e. 0, 60, 120, 180, 240 minutes).
Physical activity questionnaire | At the end of test day 1
  Questionnaire about habitual physical activity over the past 1 week. Subjects will have to report how many days per week and for how many minus they perform vigorous, moderate or relaxed physical activity.
Physical activity questionnaire | At the end of test day 2
  Questionnaire about habitual physical activity over the past 1 week. Subjects will have to report how many days per week and for how many minus they perform vigorous, moderate or relaxed physical activity.
Mood related questionnaires - The Positive and Negative Affect Schedule (PANAS scale) | At the end of test day 1
  Mood related questionnaires over the past 1 week. Subjects will have to evaluate the extent they have felt certain feelings over the past week. Score will vary between 1 (Very slightly or not at all) to 5 (Extremely).
Mood related questionnaires - The Positive and Negative Affect Schedule (PANAS scale) | At the end of test day 2
  Mood related questionnaires over the past 1 week. Subjects will have to evaluate the extent they have felt certain feelings over the past week. Score will vary between 1 (Very slightly or not at all) to 5 (Extremely).
Mood related questionnaires - Perceived Stress Scale - 10 items (PSS-10) | At the end of test day 1
  Mood related questionnaires over the past 1 week. Subjects will have to evaluate how ofter have felt certain feelings over the past week. Score will vary between 0 (Never) to 4 (Very often).
Mood related questionnaires - Perceived Stress Scale - 10 items (PSS-10) | At the end of test day 2
  Mood related questionnaires over the past 1 week. Subjects will have to evaluate how ofter have felt certain feelings over the past week. Score will vary between 0 (Never) to 4 (Very often).
Mood related questionnaires - Depression, Anxiety, Stress Scales - 21 items (DASS-21) | At the end of test day 1
  Mood related questionnaires over the past 1 week. Subjects will have to evaluate es how much the statement applied to them over the last week. Score will vary between 0 (Did not apply to me at all) to 3 (Applied to me very much or most of the time).
Mood related questionnaires - Depression, Anxiety, Stress Scales - 21 items (DASS-21) | At the end of test day 2
  Mood related questionnaires over the past 1 week. Subjects will have to evaluate es how much the statement applied to them over the last week. Score will vary between 0 (Did not apply to me at all) to 3 (Applied to me very much or most of the time).

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Verbeke, PhD, Principal Investigator — KU Leuven
Locations (2):
- Belgium (2):
  - KU Leuven/UZ Leuven, Leuven, Vlaams Brabant
  - UZ Leuven, Leuven

IPD SHARING:
Plan to Share IPD: No